CLINICAL TRIAL: NCT00301899
Title: A Phase II Study to Evaluate the Efficacy and Safety Using Combined Monoclonal Antibodies, Trastuzumab and Pertuzumab in Subjects With Her-2 Overexpressed Locally Advanced and Metastatic Breast Cancer
Brief Title: Trastuzumab and Pertuzumab in Treating Patients With Unresectable Locally Advanced or Metastatic Breast Cancer That Did Not Respond to Previous Trastuzumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 060035; 06-C-0035; NCI-P6660; CDR0000462639; NCT00263224 (obsolete NCT alias)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; male breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — pertuzumab; Trastuzumab

INTERVENTIONS:
Biological: pertuzumab
Biological: trastuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab and pertuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving trastuzumab together with pertuzumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving trastuzumab together with pertuzumab works in treating patients with unresectable locally advanced or metastatic breast cancer that did not respond to previous trastuzumab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with HER2/neu-overexpressing, inoperable locally advanced or metastatic breast cancer refractory to trastuzumab (Herceptin®)-based therapy treated with trastuzumab and pertuzumab.
* Determine the safety and tolerability of this regimen in these patients.

Secondary

* Determine the time to progression, progression-free survival, duration of response, and the percentage of patients free from disease progression at 3, 6, and 12 months.
* Correlate pre-treatment HER-2/neu phosphorylation and the phosphorylation of downstream markers of signaling pathways using tumor tissue and blood with pertuzumab sensitivity and/or trastuzumab resistance in these patients.

OUTLINE: This is an open-label study.

Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes on day 1 and pertuzumab IV over 30-60 minutes on day 2 of course 1. Beginning in course 2 and for all subsequent courses, patients receive both trastuzumab and pertuzumab on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer of 1 of the following stages:

  * Metastatic disease (stage IV)
  * Inoperable locally advanced disease

    * Disease progression after prior neoadjuvant chemotherapy required
* Disease progression on or after trastuzumab (Herceptin®) based-therapy

  * Received 1-3 prior trastuzumab-based regimens
* HER2/neu-positive tumor, defined as 3+ by fluorescent in situ hybridization
* Measurable disease, defined as at least 1 lesion that can be measured in at least one dimension
* No clinical signs or symptoms of brain and/or leptomeningeal metastases confirmed by CT scan or MRI

  * Brain and/or leptomeningeal metastases allowed if patient has stable lesions after standard treatment (surgery or radiotherapy), is asymptomatic on neurological exam, and is not receiving corticosteroid therapy to control symptoms
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Male or female
* Menopausal status not specified
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase < 5 times ULN
* AST and ALT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* LVEF above lower limit of normal by echocardiogram or MRI
* No clinical signs or symptoms of heart failure
* No uncontrolled hypertension (i.e., blood pressure ≥ 180/100 mm Hg)
* No significant valvular disease (i.e., aortic or mitral regurgitation of 3 or 4+/4+ severity or stenosis of either valve)
* No history of uncontrolled cardiac arrhythmia
* No symptomatic or asymptomatic myocardial infarction
* No angina pectoris requiring medication
* No other documented significant cardiac event
* No poorly controlled diabetes mellitus (i.e., fasting blood sugar ≥ 200 mg/dL)
* No history of hypersensitivity reaction to trastuzumab
* No AIDS
* No nonmalignant condition requiring ≥ 20 mg of prednisone (or equivalent)
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer
* No ongoing liver disease, including viral or other hepatitis, alcohol abuse, or cirrhosis
* No other serious medical illness
* No medical or psychiatric condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* More than 3 weeks since prior investigational anticancer agents
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C), major surgery, or immunotherapy
* More than 4 weeks since prior radiotherapy except short-course palliative radiotherapy for bone pain
* More than 2 weeks since prior and no concurrent oral hormonal therapy
* More than 4 weeks since prior fulvestrant
* No prior doxorubicin hydrochloride or doxorubicin HCl liposome at a cumulative dose of > 360 mg/m^2
* No prior mitoxantrone hydrochloride at a cumulative dose of > 120 mg/m^2
* No prior epirubicin hydrochloride at a cumulative dose of > 600 mg/m^2
* No prior idarubicin at a cumulative dose of > 90 mg/m^2
* No concurrent radiation therapy, including for symptomatic bone metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2005-12; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety
Minimal rate of clinical responses

SECONDARY OUTCOMES:
Time to progression
Time to response
Response duration
Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Chia Portera, MD, Study Chair — NCI - Medical Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

REFERENCES:
- [Result] Baselga J, Gelmon KA, Verma S, Wardley A, Conte P, Miles D, Bianchi G, Cortes J, McNally VA, Ross GA, Fumoleau P, Gianni L. Phase II trial of pertuzumab and trastuzumab in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer that progressed during prior trastuzumab therapy. J Clin Oncol. 2010 Mar 1;28(7):1138-44. doi: 10.1200/JCO.2009.24.2024. Epub 2010 Feb 1. PMID 20124182